CLINICAL TRIAL: NCT03914794
Title: Phase 2 Window of Opportunity Study of Pemigatinib in Non-muscle Invasive Bladder Cancer Patients With Recurrent Low- or Intermediate-Risk Tumors
Brief Title: A Study of Pemigatinib in Non-muscle Invasive Bladder Cancer Patients With Recurrent Low- or Intermediate-Risk Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J18158; IRB00194271 (Other: JHM IRB)
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer; NMIBC; Non-Muscle Invasive Bladder Cancer; Urothelial Carcinoma Recurrent
Keywords: Bladder Cancer; Non Muscle Invasive Bladder Cancer; Non-Muscle Invasive Bladder Cancer (NMIBC); NMIBC; Urothelial Carcinoma; Urothelial Cancer; Urinary Bladder Neoplasm; Bladder Neoplasm; Fibroblast inhibitors; Pemigatinib; FGFR inhibitor
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: Pemigatinib (Experimental): Patients will receive pemigatinib for 4 to 6 weeks prior to standard of care transurethral resection of bladder tumor (TURBT).
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Participants will take Pemigatinib once daily on days 1 through 28 of each cycle prior to standard of care TURBT.
  Other Names: INCB054828; FGFR inhibitor INCB054828

SUMMARY:
This phase II trial studies how well Pemigatinib (an orally administered inhibitor of fibroblast growth factor receptors 1, 2, and 3) works in non-muscle invasive bladder cancer (NMIBC) patients with recurrent tumors and a prior history of low- or intermediate-risk NMIBC tumors. Participants will receive pemigatinib for 4-6 weeks prior to standard of care transurethral resection of bladder tumor (TURBT).

DETAILED DESCRIPTION:
It is a single-arm phase 2 window of opportunity study to assess the antineoplastic activity of pemigatinib in non-muscle invasive bladder cancer (NMIBC) patients with recurrent tumors and a prior history of low- or intermediate-risk NMIBC tumors. Enrolled patients will receive pemigatinib for 4-6 weeks prior to standard of care transurethral resection of bladder tumor (TURBT). The primary endpoint will be complete response rate as determined at TURBT. Secondary endpoints will include safety profile, associations between complete response rate and tumor mutation/fusion status (e.g. FGFR3 specifically, others will also be examined) and NMIBC risk group (low- vs. intermediate-risk), and assessment of pemigatinib post-treatment urothelial tissue concentrations. The study will be conducted at 4-5 high volume bladder cancer institutions within the US and managed through the Johns Hopkins Sidney Kimmel Comprehensive Cancer Center clinical research office.

ELIGIBILITY:
Inclusion Criteria:

* Prior histologically confirmed low- or intermediate-risk non-muscle invasive urothelial carcinoma of the bladder (NMIBC) defined according to the following characteristics:

  * Low Risk

    * Initial tumor with all of the following:
    * Solitary tumor
    * Ta tumor
    * Low-grade
    * <3 cm
    * No CIS
  * Intermediate Risk

    --- All tumors not defined in the two adjacent categories (between the category of low- and high-risk)
  * High Risk

    * T1 tumor
    * High-grade
    * CIS
    * Multiple and recurrent and large (>3 cm) Ta low-grade tumors (all conditions must be met for this point on Ta low-grade tumors)
* Documented tumor recurrence as noted in standard of care follow up cystoscopy.
* ECOG (WHO) performance status 0-2
* Age ≥ 18 years old
* Patients must have the following laboratory values:

  * White blood cell count (WBC) > 3.0 K/mm3
  * Absolute neutrophil count (ANC) ≥ 1.5 K/mm3
  * Platelets ≥ 100 K/mm3
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Serum total bilirubin: ≤ 1.5 x ULN
  * ALT and AST ≤ 3.0 x ULN
  * Serum calcium < ULN
  * Serum phosphate < ULN
  * Serum creatinine ≤ 1.5 x ULN or serum creatinine > 1.5 - 3 x ULN if calculated creatinine clearance (CrCl) is ≥ 30 mL/min using the modified Cockcroft-Gault equation
* Patients who give a written informed consent obtained according to local guidelines

Exclusion Criteria:

* Patients with concurrent upper urinary tract (i.e. ureter, renal pelvis) non-invasive urothelial carcinoma.
* Patients with high grade urothelial carcinoma on their most recent urine cytology.
* Patients with another active second malignancy other than non-melanoma skin cancers and biochemical relapsed prostate cancer. (Patients that have completed all necessary therapy and are considered to be at less than 30% risk of relapse are not considered to have an active second malignancy and are eligible for enrollment.)
* Patients who have received the last administration of an anti-cancer therapy including chemotherapy, immunotherapy, and monoclonal antibodies ≤ 4 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have received prior selective fibroblast growth factor receptor targeting agents (i.e. pemigatinib, dovitinib, BGJ398, AZD4547, JNJ-42756493, etc.).
* Patients who have had radiotherapy ≤ 4 weeks prior to starting study drug, or who have not recovered from radiotherapy toxicities
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures (i.e. TURBT), percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Complete response rate of pemigatinib therapy | 6 weeks
  The number of participants with a complete response to pemigatinib therapy. Tumor complete response is defined as the complete absence of any stage bladder tumor on post-treatment Transurethral Resection of a Bladder Tumor (TURBT) and no evidence of recurrent urothelial carcinoma on post-treatment urine cytology.

SECONDARY OUTCOMES:
Characterize the safety profile of pemigatinib therapy | 4 years
  Number of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 toxicities
Number of Participants with Complete Response and FGFR3 Mutational Status | Up to 4 weeks
Number of Participants with Non-Muscle Invasive Bladder Cancer (NMIBC) and Complete Response | Up to 4 years
  Number of participants with complete response rate and baseline NMIBC risk group (low- vs. intermediate-risk)
Maximal concentration (Cmax, nmol/L) of pemigatinib in urothelial tissue at post-treatment TURBT | Up to 4 weeks
Relapse Free Survival (RFS) at 6 months | 6 months
  Number of months from achieving a complete response at initial post-treatment TURBT until relapse.
Relapse Free Survival (RFS) at 12 months | 12 months
  Number of months from achieving a complete response at initial post-treatment TURBT until relapse.
Relapse Free Survival (RFS) at 24 months | 24 months
  Number of months from achieving a complete response at initial post-treatment TURBT until relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Noah M Hahn, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (6):
- United States (6):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Associated Medical Professionals Urology, Syracuse, New York
  - Midlantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No